CLINICAL TRIAL: NCT04515563
Title: Effectiveness of Different Exercise Intensities and Frequencies of Walking Exercise on Improving Cognitive Function in Older Adults With Mild Cognitive Impairment: a Pilot Randomized Controlled Trial
Brief Title: Effectiveness of Walking Exercise in Improving Cognitive Function in Older Adults With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Parco M. Siu, PhD, Associate Professor & Division Head, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-3030059835-007
Record Dates: First submitted 2020-08-10; First posted 2020-08-17 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Mild Cognitive Impairment
Keywords: Aerobic exercise; Walking exercise; Mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control Group (Placebo Comparator): Subjects in the care control group will perform once-a-week stretching exercise intervention. Each session lasts for 75 minutes and covers the major muscle groups.
  Interventions: Behavioral: Stretching exercise
- Low-frequency, moderate-intensity walking group (Experimental): A personalized walking exercise program will be arranged and conducted individually. Exercise training will be prescribed as a 12-week program, with one 150-minute instructor-led session per week. In each session, there will be 5-min warm-up and cool-down, and 150 minutes of exercise time. If needed, there will be two 10-20 min breaks for the subject to get hydrated and rest. The intensity level will be set to 3.5 metabolic equivalents (METs), in which 1 MET refers to the metabolic rate during quiet sitting [23]. During the training session, the heart rate will be continuously monitored by Polar E68 HR Sensor to make sure the subject meet the exercise intensity. 10 bpm fluctuation of the heart rate is acceptable [24].
  Interventions: Behavioral: Low-frequency, moderate-intensity walking group
- High-frequency, moderate-intensity walking group (Experimental): Intervention of high-frequency, moderate-intensity walking exercise will be given to subjects in this group. A personalized walking exercise program will be arranged and conducted individually. Exercise training will be prescribed as a 12-week program, with three 50-minute instructor-led sessions per week. In each session, there will be 5-min warm-up and cool-down, and 50 minutes of exercise time. If needed, there will be one 10-20 min break for the subject to get hydrated and rest. The intensity level will be set to 3.5 metabolic equivalents (METs), in which 1 MET refers to the metabolic rate during quiet sitting [23]. During the training session, the heart rate will be continuously monitored by Polar E68 HR Sensor to make sure the subject meet the exercise intensity. 10 bpm fluctuation of the heart rate is acceptable [24].
  Interventions: Behavioral: High-frequency, moderate-intensity walking group
- Low-frequency, vigorous-intensity walking group (Experimental): Intervention of low-frequency, vigorous-intensity walking exercise will be given to subjects in this group. A personalized walking exercise program will be arranged and conducted individually. Exercise training will be prescribed as a 12-week program, with one 75-minute instructor-led session per week. In each session, there will be 5-min warm-up and cool-down, and 75 minutes of exercise time. If needed, there will be two 10-20 min breaks for the subject to get hydrated and rest. The intensity level will be set to 7.0 metabolic equivalents (METs), in which 1 MET refers to the metabolic rate during quiet sitting [23]. During the training session, the heart rate will be continuously monitored by Polar E68 HR Sensor to make sure the subject meet the exercise intensity. 10 bpm fluctuation of the heart rate is acceptable [24].
  Interventions: Behavioral: Low-frequency, vigorous-intensity walking group
- High-frequency, vigorous-intensity walking group (Experimental): Intervention of high-frequency, vigorous-intensity walking exercise will be given to subjects in this group. A personalized walking exercise program will be arranged and conducted individually. Exercise training will be prescribed as a 12-week program, with three 25-minute instructor-led sessions per week. In each session, there will be 5-min warm-up and cool-down, and 25 minutes of exercise time. If needed, there will be a 10-20 min break for the subject to get hydrated and rest. The intensity level will be set to 7.0 metabolic equivalents (METs), in which 1 MET refers to the metabolic rate during quiet sitting [23]. During the training session, the heart rate will be continuously monitored by Polar E68 HR Sensor to make sure the subject meet the exercise intensity. 10 bpm fluctuation of the heart rate is acceptable [24].
  Interventions: Behavioral: High-frequency, vigorous-intensity walking group

INTERVENTIONS:
Behavioral: Stretching exercise — Control Group
  Arms: Control Group
Behavioral: Low-frequency, moderate-intensity walking group — once-a-week walking exercise at moderate intensity
  Arms: Low-frequency, moderate-intensity walking group
Behavioral: High-frequency, moderate-intensity walking group — thrice-a-week walking exercise at moderate intensity
  Arms: High-frequency, moderate-intensity walking group
Behavioral: Low-frequency, vigorous-intensity walking group — once-a-week walking exercise at vigorous intensity
  Arms: Low-frequency, vigorous-intensity walking group
Behavioral: High-frequency, vigorous-intensity walking group — thrice-a-week walking exercise at vigorous intensity
  Arms: High-frequency, vigorous-intensity walking group

SUMMARY:
The increasing prevalence of mild cognitive impairment (MCI) in our rapidly aging population prompts the need for devising effective interventions to prevent the onset of cognitive impairment and delay its progression to dementia. The benefits of aerobic exercise on the cognitive function in older adults with MCI are well-documented. However, exercise protocols and outcome measurement tools in the current literature are highly heterogeneous. It is therefore imperative to develop standard exercise prescription protocol for the MCI population or to examine the effectiveness of the existing, well-established exercise guidelines. The World Health Organization (WHO) recommends adults (18 - 64 years of age) and older adults (65 years and older) to perform 150 minutes of moderate-intensity or 75 minutes of vigorous-intensity aerobic physical activity per week to improve cardiorespiratory and muscular fitness, bone health, and reduce the risk of non-communicable diseases and depression. Nonetheless, few studies have determined the effectiveness of the WHO Global Recommendations on Physical Activity for Health guideline in improving cognitive function in older adults with MCI. This study thus aims to evaluate the effectiveness of the WHO Physical Activity Recommendations in improving cognitive function in older adults with MCI. In 2017, the American Academy of Neurology (AAN) updated the Practice Guideline for Mild Cognitive Impairment, in which they recommended patients diagnosed with MCI to perform exercise at least twice a week for at least 6 months to gain cognitive benefits. This recommendation was based on two class-II studies, in which a 6-month twice-a-week 90-minute multicomponent exercise program helped maintain global cognition, and selective attention improved significantly following a 6-month twice-a-week 60-minute multicomponent exercise program. While they provided pivotal insights into clinical practice, there were several limitations for these two studies. For instance, in the study conducted by Nagamatsu et al., only female subjects were recruited, and therefore lead to low generalizability. These two studies focused on multi-component exercise intervention which included resistance training, aerobic training, and balance training, and the duration of each component was short (around 20 - 30 minutes). Studies that focus on single exercise modality with longer session duration are warranted to unveil the efficacy of a certain exercise modality in improving cognitive function. In this study, we will evaluate the effectiveness of aerobic exercise on improving cognitive function in older adults with MCI. We intend to follow the WHO Recommendations, focusing on evaluating the effect of different exercise intensities (moderate versus vigorous) and frequencies (once versus thrice per week) of aerobic exercise on improving the cognitive function in older adults with mild cognitive impairment. In particular, the AAN also suggested that physical activity of at least twice a week is necessary to produce cognitive benefits. We, therefore, aim to investigate whether one session per week would also suffice to improve the cognitive function in older adults with MCI.

Aims: To examine the effectiveness of 12-week WHO Global Recommendations on Physical Activity for Health in practice in improving the cognitive function in older adults with MCI.

ELIGIBILITY:
Inclusion Criteria:

1. Older adults aged ≥ 50 years old;
2. Ethnic Chinese;
3. Diagnosed with mild cognitive impairment (MCI) under the Mayo Clinic criteria [8-10]: 1). Subjective complaint about a decline in cognitive function; 2). Total score in the Hong Kong version of the Montreal Cognitive Assessment is below the 7th percentile of the age- and education-corrected normative data of Hong Kong; 3). The decline in cognitive function does not impair daily functioning, as revealed by getting ≥ 2 marks in every item on the Chinese Lawton Instrumental Activities of Daily Living Scale (4-point Scale).

Exclusion Criteria:

1. Diagnosis of dementia/Alzheimer's disease, or currently using antidementia medication;
2. Incapable of participating in physical exercise with major confounding conditions that are known to affect mobility. Specifically designed questionnaires will be used to screen for exclusion criteria including 1). Cannot walk without assistive device; 2). Any serious somatic condition that prevents walking exercise participation.
3. History of major diseases e.g. cancer, cardio-/cerebrovascular, neurodegenerative and renal diseases;
4. Diagnosis of psychiatric diseases, or currently using psychiatric medication.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Global cognition-Hong Kong Montreal Cognitive Assessment (HK-MoCA) score | 3-month follow-up
  Age- and education-corrected Hong Kong Montreal Cognitive Assessment (HK-MoCA). The HK-MoCA is a validated assessment for cognitive screening that takes into account different domains of cognition, which will enable the researchers to achieve a better understanding of the global cognitive profile of the individual. Higher score indicates better global cognitive performance.

SECONDARY OUTCOMES:
Objective cognitive score | 3-month follow-up
  The NIH Toolbox Cognitive Function Battery (CFB) will be used to evaluate the various cognitive domains [15]. CFB will be delivered on a tablet computer. A total objective cognitive score will be generated, while a higher score indicates better cognitive performance.
Working memory-Digit Span test | 3-month follow-up
  Working memory will be measured by Digit Span test in paper-pencil based manner. Higher score indicates better cognitive performance.
Working memory-Verbal Fluency Test | 3-month follow-up
  Verbal Fluency Test will be used to measure working memory. Higher score indicates better cognitive performance.
Executive function-Stroop test | 3-month follow-up
  Executive function will be measured by Stroop test. Shorter completion time indicates better performance.
Executive function-Trail Making test | 3-month follow-up
  Executive function will be measured by Trail Making test. Shorter completion time indicates better performance.
Subjective cognitive report | 3-month follow-up
  Cognitive self-report questionnaire (CSQR) will be used to test the subjective cognitive performance. CSQR is validated in HK and consists of 20 questions with overall score ranging from 0-100. Higher score indicates worse self-perception on cognitive performance.
Remission rate-Chinese Abbreviated Mild Cognitive Impairment Test (CAMCI) | 3-month follow-up
  Chinese Abbreviated Mild Cognitive Impairment Test (CAMCI) will be used to classify participants into MCI and non-MCI category. The remission rate will be calculated as remission rate = number of participants in non-MCI category / number of total participants.
Remission rate-Hong Kong Montreal Cognitive Assessment (HK-MoCA) | 3-month follow-up
  Age- and education-corrected Hong Kong Montreal Cognitive Assessment (HK-MoCA). The HK-MoCA is a validated assessment for cognitive screening that takes into account different domains of cognition, which will enable the researchers to achieve a better understanding of the cognitive profile of the individual. MoCA will be used to classify participants into MCI and non-MCI category. The remission rate will be calculated as remission rate = number of participants in non-MCI category / number of total participants.
VO2max | 3-month follow-up
  A VO2max test will be conducted using a calibrated motor-driven treadmill by continuous metabolic VO2 measurement using a COSMED Quark Series telemetric gas analysis system. The test will be performed using a modified bruce protocol. VO2, Borg's rating of perceived exertion (RPE) and heart rate (HR) will be continuously recorded. The maximal attainable heart rate will be recorded as the peak heart rate (HRpeak).
Body fat mass | 3-month follow-up
  Body fat mass of participants will be measured by dual-energy X-ray absorptiometry (DXA).
Lean mass | 3-month follow-up
  Lean mass of participants will be measured by dual-energy X-ray absorptiometry (DXA).
Bone mineral density | 3-month follow-up
  Bone mineral density of participants will be measured by dual-energy X-ray absorptiometry (DXA).
Habitual sleep | 3-month follow-up
  The Pittsburgh Sleep Quality Index (PSQI) is a standardized instrument to estimate sleep quantity and quality. The PSQI has been commonly used to distinguish people with primary insomnia from normal sleepers. The Chinese version of PSQI has been validated to have a satisfactory Cronbach's alpha of 0.82-0.83 and test-retest reliability of 0.85 among Hong Kong Chinese older adults. The overall score ranges from 0 to 24 while a higher score indicates worse sleep quality.
Quality of Life-12-item Short Form Survey (SF-12) | 3-month follow-up
  The 12-item Short Form Survey (SF-12) will be used to assess the quality of life of the participant and higher scores (physical and mental sub-scale) indicate better quality of life.
Depression level | 3-month follow-up
  Patient Health Questionnaire-9 (PHQ-9) will also be used to assess the mental health of the subjects. A PHQ-9 score of ≥ 10 has a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 correspond to mild, moderate, moderately severe, and severe depression, respectively. Results are similar in the primary care and obstetrics-gynecology samples. The PHQ-9 is a reliable and valid measure of depression severity and its brevity make the PHQ-9 a useful clinical and research tool.
Mental health | 3-month follow-up
  Hospital Anxiety and Depression Scale (HADS) will used to measure the mental health of participants. It is a 7-item questionnaire having an overall score that ranges from 0 to 21 (with sub-scales for both anxiety and depression), with a higher score indicating more severe symptoms.
Anxiety level | 3-month follow-up
  Generalized Anxiety Disorder 7-item (GAD-7) scale will be used to measure the anxiety level of participants. It is a 7-item questionnaire having an overall score that ranges from 0 to 21 with a higher score indicating more severe symptoms.
Physical activity | 3-month follow-up
  The International Physical Activity Questionnaire (IPAQ) will be used to assess the activity level of the subjects.
Balance performance | 3-month follow-up
  The balance ability of the subjects will be measured by single leg standing test. The longer standing duration indicates better balance performance.

CONTACTS AND LOCATIONS:
Overall Officials: MING FAI SIU, Ph.D., Study Director — School of Public Health, the University of Hong Kong
Locations (1):
- Li Kai Shing Faculty of Medicine, Hong Kong, Southern District, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data of individual participants that underlie the results reported in this trial, after de-identification including text, tables, figures, and appendices, as well as study protocol and statistical analysis plan, will be shared after 3 months of study publication. Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for the data requests, a data-access agreement needs to be signed.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months after study publication and ending 3 years.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for the data requests, a data-access agreement needs to be signed.

REFERENCES:
- [Derived] Yu DJ, Yu AP, Bernal JDK, Fong DY, Chan DKC, Cheng CP, Siu PM. Effects of exercise intensity and frequency on improving cognitive performance in middle-aged and older adults with mild cognitive impairment: A pilot randomized controlled trial on the minimum physical activity recommendation from WHO. Front Physiol. 2022 Sep 19;13:1021428. doi: 10.3389/fphys.2022.1021428. eCollection 2022. PMID 36200056